CLINICAL TRIAL: NCT05444608
Title: Evaluation of the Effect of Use of Breast Milk Odor and White Noise on Pain Management During Heel Lance in Premature Newborns: A Randomized Controlled Study
Brief Title: Premature Newborn Pain Management: The Effects of Breast Milk Odor and White Noise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Burcu Otlu, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AnkaraU06BO
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pain
Keywords: Newborn; Pain; Breast milk odor; White noise; Heel lance
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This randomized controlled experimental study will performing to investigate the effect of smelling breast milk and listening to white noise in reducing pain during heel puncture
Who Masked: Participant, Outcomes Assessor
Masking Description: A sponge soaked in saline was placed next to the babies listening to white noise, and a non-working loudspeaker was placed on the toe of the babies who smelled breast milk. The assessment was made by academics other than the researcher by muting the video recordings. The babies were considered blind because they did not know which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Data will be collected during heel blood sampling for blood sugar control from newborns randomly assigned to the control group. Babies in the control group will not be allowed to smell breast milk or listen to white noise.The newborn in the control group will continue to receive routine care.Camera recording will start 5 minutes before the procedure and lasting 5 minutes after the procedure.
- Breast Milk Odor Group (Experimental): Data will be collected during heel blood sampling for blood sugar control from newborns randomly assigned to the breast milk odor group.Before the intervention, 2 ml of breast milk will be dripped into sterile sponge and the sponge will be placed within 3 cm of the newborn's nose.Babies in this group will start to smell their mother's milk 5 minutes before the procedure and will continue to smell for 5 minutes after the procedure.Camera recording will start 5 minutes before the procedure and lasting 5 minutes after the procedure.
  Interventions: Behavioral: Breast milk olfactory stimulation
- White Noise Group (Experimental): Data will be collected during heel blood sampling for blood sugar control from newborns randomly assigned to the white noise listening group.Before the intervention , a bluetooth speaker will be placed at the baby's feet. The speaker will be connected to the phone and the sound level will be adjusted to 50 decibels by means of a decibel meter. The baby will be started to listen to white noise 5 minutes before the procedure.Camera recording will start 5 minutes before the procedure and lasting 5 minutes after the procedure.
  Interventions: Behavioral: White noise auditory stimulation

INTERVENTIONS:
Behavioral: Breast milk olfactory stimulation — Before the intervention, 2 ml of breast milk will be dripped into sterile sponge and the sponge will be placed within 3 cm of the newborn's nose.Babies in this group will start to smell their mother's milk 5 minutes before the procedure and will continue to smell for 5 minutes after the procedure.
  Arms: Breast Milk Odor Group
Behavioral: White noise auditory stimulation — Before the intervention, a bluetooth speaker will be placed at the baby's feet. The speaker will be connected to the phone and the sound level will be adjusted to 50 decibels by means of a decibel meter. The baby will be started to listen to white noise 5 minutes before the procedure and will continue to listen for 5 minutes after the procedure.
  Arms: White Noise Group

SUMMARY:
This study will conduct to evaluate the effect of using white noise and breast milk odor on pain during heel lance procedure in premature newborns. This study is a randomized controlled trial.

The study will conduct with premature newborns who were born between 34 and 37 weeks of gestation. The premature newborns will be divided into three groups by application of pain relief methods during heel lance to check blood sugar in newborns. These groups can be described as breast milk odor (n=22), white noise (n=22) and control group (n=22). The intervention will start 5 minutes before the procedure and last 5 minutes after the procedure. The infants will be recorded with a video camera by researcher before, during, and after the procedure. Premature Infant Pain Profile Revised (PIPP-R) will be used for pain grading.

DETAILED DESCRIPTION:
The sense of pain develops in infants after the 20th gestational weeks with the initiation of communication between the cortex and the thalamus. Babies in the newborn period can respond physiologically, behaviorally and hormonal to painful stimuli which they experienced. Responses that emerge as a result of pain experience may adversely affect the current state of the newborn and its growth and development in the long term. One of the painful procedures that the newborn is frequently exposed to at the beginning of the extra-uterine life is blood collection from the heel. Pharmacological and non-pharmacological methods can be applied to alleviate the pain sensation experienced by newborns during these procedures. The existence of possible side effects of pharmacological methods has led to need to use non-pharmacological methods more effectively. In this study, it was aimed to investigate the effectiveness of breast milk odor and white noise, which are non-pharmacological methods, to the pain caused by heel puncture.

Main hypothesizes of the study can be listed as:

H11: Breast milk smelling during heel lancing in preterm newborn infants effectively reduces the infant's procedure-related pain.

H01: Breast milk smelling during heel lancing in preterm newborn infants is not effective in reducing the procedure-related pain of the infant.

H12: Listening to white noise during heel lancing in preterm newborn babies effectively reduces the baby's procedure-related pain.

H02: Listening to white noise during heel lancing in preterm newborn infants is not effective in reducing the procedure-related pain of the infant.

H13: Breast milk smelling during heel puncture in preterm newborn infants is more effective than white noise in reducing the procedure-related pain of the infant.

H03: Breast milk smelling during heel puncture in preterm newborn infants is not more effective than white noise in reducing the procedure-related pain of the infant.

H14: Listening to white noise during heel lancing in preterm newborn babies is more effective than breast milk odor in reducing the procedure-related pain of the baby.

H04: Listening to white noise during heel lancing in preterm newborn babies is not more effective than breast milk odor in reducing the procedure-related pain of the infant.

The population of the study will consist of preterm babies born between 34-37 weeks of gestation, who were hospitalized in the Neonatal Intensive Care Unit mother-baby room, and postnatal service of Ankara University Faculty of Medicine, Cebeci Application and Research Hospital, between May 2022 and October 2022 and for whom heel blood sampling is requested.The sample of the study will consist of 66 (white noise=22, breast milk odor=22, control=22) infants who met the case selection criteria and were randomly assigned to groups. Babies will be made to listen to white noise or smell breast milk for 5 minutes before the heel blood collection procedure, during the procedure and 5 minutes after the procedure in accordance with the group they are involved. Only routine nursing care will be applied to the control group, no additional intervention. All the infants in three different groups will be recorded by video camera. Recording will start 5 minutes before the heel lance procedure and continue during the procedure and 5 minutes after the procedure. Pain assessments will be made by another researcher through video recordings. Newborns pain will evaluate with the PIPP-R pain scale 5 minutes before procedure (at the beginnings of intervention), 2 minutes before procedure, at the time of the procedure and 5 minutes after the procedure. Heart rate and oxygen saturation will be recorded at the same times.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 34 and 37 weeks
* birth weight over 1500 g
* Taking blood from the heel for the purpose of measuring blood sugar
* Starting feeding with breast milk
* Parental consent

Exclusion Criteria:

* Having a chromosomal abnormality
* Presence of neonatal seizures
* Presence of intracranial bleeding (grade III-IV)
* Presence of craniofacial malformation
* Presence of congenital hearing loss
* Babies with perinatal asphyxia
* Babies using sedatives, muscle relaxants and antiepileptics
* Babies whose mothers have a history of substance use

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Pain | up to 7 days
  Premature Infant Pain Profile-Revised
  The scale includes seven criteria. Facial expressions (frown, squint, prominence of the nasolabial groove) represent three criteria. Two additional criteria are changes in heart rate and reduction in oxygen saturation. The remaining criteria are gestational week and behavioral status (active-awake, quiet-wake, active-asleep and quiet-sleeping). According to the scale, the highest score is 21 for prematures and 18 for term newborns. According to the scale scoring, 0-6 points indicate mild pain, 7-12 points moderate pain, and 13-21 points severe pain in a premature baby.
Physiological Findings | up to 7 days
  Physiological Findings Follow-up Chart

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Akcan E, Polat S. Comparative Effect of the Smells of Amniotic Fluid, Breast Milk, and Lavender on Newborns' Pain During Heel Lance. Breastfeed Med. 2016 Aug;11(6):309-314. doi: 10.1089/bfm.2015.0174. Epub 2016 Jun 17. PMID 27315487
- [Background] Alemdar DK. Effect of recorded maternal voice, breast milk odor, and incubator cover on pain and comfort during peripheral cannulation in preterm infants. Appl Nurs Res. 2018 Apr;40:1-6. doi: 10.1016/j.apnr.2017.12.001. Epub 2017 Dec 14. PMID 29579482
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn; American Academy of Pediatrics Section on Surgery; Canadian Paediatric Society Fetus and Newborn Committee; Batton DG, Barrington KJ, Wallman C. Prevention and management of pain in the neonate: an update. Pediatrics. 2006 Nov;118(5):2231-41. doi: 10.1542/peds.2006-2277. PMID 17079598
- [Background] Baudesson de Chanville A, Brevaut-Malaty V, Garbi A, Tosello B, Baumstarck K, Gire C. Analgesic Effect of Maternal Human Milk Odor on Premature Neonates: A Randomized Controlled Trial. J Hum Lact. 2017 May;33(2):300-308. doi: 10.1177/0890334417693225. Epub 2017 Mar 27. PMID 28346843
- [Background] Brummelte S, Grunau RE, Chau V, Poskitt KJ, Brant R, Vinall J, Gover A, Synnes AR, Miller SP. Procedural pain and brain development in premature newborns. Ann Neurol. 2012 Mar;71(3):385-96. doi: 10.1002/ana.22267. Epub 2012 Feb 28. PMID 22374882
- [Background] Cakirli M, Acikgoz A. A Randomized Controlled Trial: The Effect of Own Mother's Breast Milk Odor and Another Mother's Breast Milk Odor on Pain Level of Newborn Infants. Breastfeed Med. 2021 Jan;16(1):75-81. doi: 10.1089/bfm.2020.0222. Epub 2020 Oct 20. PMID 33085532
- [Background] Cetinkaya S, Yavas Celik M, Ozdemir S. Effect of white noise on alleviating the pain of new-born during invasive procedures. J Matern Fetal Neonatal Med. 2022 Apr;35(8):1426-1432. doi: 10.1080/14767058.2020.1755652. Epub 2020 Apr 21. PMID 32316794
- [Background] Cignacco E, Hamers JP, Stoffel L, van Lingen RA, Gessler P, McDougall J, Nelle M. The efficacy of non-pharmacological interventions in the management of procedural pain in preterm and term neonates. A systematic literature review. Eur J Pain. 2007 Feb;11(2):139-52. doi: 10.1016/j.ejpain.2006.02.010. Epub 2006 Apr 3. PMID 16580851
- [Background] Doesburg SM, Chau CM, Cheung TPL, Moiseev A, Ribary U, Herdman AT, Miller SP, Cepeda IL, Synnes A, Grunau RE. Neonatal pain-related stress, functional cortical activity and visual-perceptual abilities in school-age children born at extremely low gestational age. Pain. 2013 Oct;154(10):1946-1952. doi: 10.1016/j.pain.2013.04.009. Epub 2013 Apr 8. PMID 23711638
- [Background] Dora O, Buyuk ET. RETRACTED: Effect of White Noise and Lullabies on Pain and Vital Signs in Invasive Interventions Applied to Premature Babies. Pain Manag Nurs. 2021 Dec;22(6):724-729. doi: 10.1016/j.pmn.2021.05.005. Epub 2021 Jun 28. PMID 34210600
- [Background] Grunau RE, Holsti L, Peters JW. Long-term consequences of pain in human neonates. Semin Fetal Neonatal Med. 2006 Aug;11(4):268-75. doi: 10.1016/j.siny.2006.02.007. Epub 2006 Apr 24. PMID 16632415
- [Background] Kahraman A, Gumus M, Akar M, Sipahi M, Bal Yilmaz H, Basbakkal Z. The effects of auditory interventions on pain and comfort in premature newborns in the neonatal intensive care unit; a randomised controlled trial. Intensive Crit Care Nurs. 2020 Dec;61:102904. doi: 10.1016/j.iccn.2020.102904. Epub 2020 Jul 9. PMID 32653359
- [Background] Kucuk Alemdar D, Kardas Ozdemir F. Effects of Having Preterm Infants Smell Amniotic Fluid, Mother's Milk, and Mother's Odor During Heel Stick Procedure on Pain, Physiological Parameters, and Crying Duration. Breastfeed Med. 2017 Jun;12:297-304. doi: 10.1089/bfm.2017.0006. Epub 2017 Apr 17. PMID 28414516
- [Background] Maayan-Metzger A, Kedem-Friedrich P, Bransburg Zabary S, Morag I, Hemi R, Kanety H, Strauss T. The Impact of Preterm Infants' Continuous Exposure to Breast Milk Odor on Stress Parameters: A Pilot Study. Breastfeed Med. 2018 Apr;13(3):211-214. doi: 10.1089/bfm.2017.0188. Epub 2018 Mar 12. PMID 29620936
- [Background] Rad ZA, Aziznejadroshan P, Amiri AS, Ahangar HG, Valizadehchari Z. The effect of inhaling mother's breast milk odor on the behavioral responses to pain caused by hepatitis B vaccine in preterm infants: a randomized clinical trial. BMC Pediatr. 2021 Feb 1;21(1):61. doi: 10.1186/s12887-021-02519-0. PMID 33522927
- [Background] Stevens BJ, Gibbins S, Yamada J, Dionne K, Lee G, Johnston C, Taddio A. The premature infant pain profile-revised (PIPP-R): initial validation and feasibility. Clin J Pain. 2014 Mar;30(3):238-43. doi: 10.1097/AJP.0b013e3182906aed. PMID 24503979
- [Background] Taddio A, Shah V, Atenafu E, Katz J. Influence of repeated painful procedures and sucrose analgesia on the development of hyperalgesia in newborn infants. Pain. 2009 Jul;144(1-2):43-8. doi: 10.1016/j.pain.2009.02.012. Epub 2009 Mar 28. PMID 19329255
- [Background] Taplak AS, Bayat M. Psychometric Testing of the Turkish Version of the Premature Infant Pain Profile Revised-PIPP-R. J Pediatr Nurs. 2019 Sep-Oct;48:e49-e55. doi: 10.1016/j.pedn.2019.06.007. Epub 2019 Jun 19. PMID 31229348
- [Derived] Otlu B, Esenay FI. Use of Mothers Milk Odor and White Noise on Pain Management in Preterm Infants: A Randomized Controlled Trial. Adv Neonatal Care. 2025 Feb 1;25(1):28-36. doi: 10.1097/ANC.0000000000001214. Epub 2024 Dec 16. PMID 39681072